CLINICAL TRIAL: NCT00528346
Title: Treatment Of Chronic Pain Using Real-time Functional MRI Trial
Brief Title: Treatment Of Chronic Pain Using Real Time fMRI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Omneuron (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Christopher deCharms, Principal Investigator, Omneuron
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2R44NS050642-06 (NIH)
Record Dates: First submitted 2007-09-11; First posted 2007-09-12 (Estimated); Last update posted 2011-04-26 (Estimated); Status verified 2011-04

CONDITIONS: Chronic Pain
Keywords: chronic pain; functional magnetic resonance imaging; fMRI; cognitive training
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Participants will see their own brain activation.
  Interventions: Behavioral: cognitive training using fMRI
- 2 (Placebo Comparator): Participants will see simulated data that does not come from their own brains.
  Interventions: Behavioral: placebo

INTERVENTIONS:
Behavioral: cognitive training using fMRI — Participants will be scanned using fMRI while they employ the cognitive training strategies-allowing them to view their brain activity.
  Arms: 1
Behavioral: placebo — Some participants will see simulated data that does not come from their own brains.
  Arms: 2

SUMMARY:
The purpose of this study is to test a new investigational method for treatment of chronic pain using cognitive training guided by functional magnetic resonance imaging (fMRI).

DETAILED DESCRIPTION:
Chronic pain is a substantial medical and economic problem, and is often unresponsive to conventional treatment. In this study, scientists will seek to decrease pain by increasing control over pain using newly-developed brain imaging methods to train people to control their own brain activation. This is the first clinical application of a recently-developed technology allowing a person to watch their own brain activation second-by-second and to learn to control it. It may provide a means to train people to control chronic pain by controlling their own brain states.

The purpose of the study is to evaluate real-time functional magnetic resonance imaging (fMRI) feedback for treating chronic pain diagnoses, including fibromyalgia, neuralgia, neuropathy, migraine, and complex regional pain syndrome (CRPS)/reflex sympathetic dystrophy (RSD). The study will also measure the impact of cognitive training for pain control on activations from the areas of the brain involved in pain.

All participants in this study will receive a new form of cognitive training for controlling pain. Participants will be scanned using fMRI while they employ the cognitive training strategies-allowing them to view their brain activity. Some participants will see their own brain activation during this process while other participants will see very similar but simulated data that does not come from their own brains.

Participation in the study will last about 6 months with 12 visits that includes 6 sessions in an MRI scanner. Recruitment for this trial is limited to persons in the San Francisco Bay area. Participants must be able to attend sessions in Menlo Park, CA. Participants will be reimbursed for travel time within the Bay area.

Information gained from this study may help in developing potential future treatments for chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed chronic pain. Some example diagnoses include: CRPS, RSD, neuropathy, neuralgia, fibromyalgia, or migraine.
* No implanted medical devices that are not compatible with MRI (spinal cord stimulator/pump, pacemaker, surgical aneurysm clip, etc)
* No recent history of severe psychiatric illness
* Weight less than 220 lbs.
* Able to be scanned in MRI without claustrophobia
* No facial tattoos, non-removable metal implants, piercings, or extensive dental work.
* Not pregnant or having fertility treatments

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2007-09; Primary Completion 2011-08 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Measures of Pain Magnitude; McGill Pain Questionnaire; Visual Analogue Scale; Coping Strategies; Pain Catastrophizing Scale; Beck Depression Inventory; Treatment Outcome of Pain States; Increased control over brain activation measured using fMRI | duration of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Christopher deCharms, PhD, Principal Investigator — Omneuron
Locations (1):
- Omneuron, 99 El Camino Real, Menlo Park, California, United States